CLINICAL TRIAL: NCT03627897
Title: Erector Spinae Plane Block for Postoperative Analgesia in Pediatric Patients Undergoing Cardiac Surgery: A Double-Blind, Randomized, Controlled Study
Brief Title: ESP Block in Pediatric Patients for Postoperative Analgesia
Acronym: ESP1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Principal investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESPediatrics
Record Dates: First submitted 2018-08-04; First posted 2018-08-14 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Opioid Use; Pain, Postoperative; Quality of Life
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The children will randomly assigned into two study groups by a computer-generated random number list. The children in group B will be administered bilateral ESPB with 0.25% bupivacaine by non-blinded researcher to the study groups), while the children in group C will be not administered any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional analgesia group (Experimental): ESP block at bilateral side will be performed in the lateral decubitis position and at T5 transverse process level by using 10-MHz liner ultrasound probe. The probe will be located 1 cm lateral to T5 spinous process in longitudinal parasagittal orientation. Simplex A 50mm (B.Braun, Germany) will be inserted by using out of plane technique. The ESP blocks proceed with 0,5 ml/kg of 0,25% bupivacaine
  Interventions: Drug: Bupivacain
- Control group (Other)
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Bupivacain — The erector spinae plane blocks proceed with 0,5 ml/kg of 0,25% bupivacain (Group B).
  Arms: Regional analgesia group
Drug: saline — No drugs or interventions were administered to the control group.
  Arms: Control group

SUMMARY:
Pediatric cardiac surgery is associated with moderate to severe postoperative pain that is related to median sternotomy. In a fast-track protocol, used in modern-day cardiac surgical care, early extubation may be facilitated by effective postoperative pain control, which also helps in maintaining hemodynamic stability This prospective, randomized, and double-blind study is designed to examine the efficacy and safety of the ESP block on the postoperative analgesia in pediatric patients after cardiac surgery.

40 pediatric patients aged 2-10 years, undergoing cardiac surgery with median sternotomy will be enrolled. Children received oral premedication of midazolam 0.5 mg/kg. After i.v. access will be obtained, fentanyl 5 µg/kg will be given. Anesthesia will be induced with 2-3 mg/kg propofol and all children will receive rocuronium 0,6 mg/kg for tracheal intubation.Subsequently, fentanyl 5 µg/kg will be administered prior to incision and an additional 5 microg/kg of fentanyl given prior to CPB. Anesthesia will be maintained with %2-3 sevoflurane. Fentanyl 1 µg/kg will be given before skin closure at the end of surgery. Patients were randomly assigned to a study group by the computer generated number table. Children in group B were administered bilateral ESPB with 0.25% bupivacaine, while children in group C did not receive any intervention. Following inhalational induction and endotracheal tube placement, the patient will be turned into a left lateral decubitus position and bilateral ESP block will be performed under aseptic conditions.

ESP block at bilateral side will be performed in the lateral decubitis position and at T5 transverse process level by using 10-MHz liner ultrasound probe. The probe will be located 1 cm lateral to T5 spinous process in longitudinal parasagittal orientation. Simplex A 50mm (B.Braun, Germany) will be inserted by using out of plane technique. The ESP blocks proceed with 0,5 ml/kg of 0,25% bupivacaine (Group B).

Postoperative care: All the patients then will be shifted to the intensive care unit (ICU) after the surgery and managed with the institution's ICU protocol for postoperative pain management and ventilation.The postoperative analgesia will be provided with rescue intravenous (IV) morphine 0.05 mg/kg. Both the groups will receive IV paracetamol 15 mg/kg every 6 hours as a component of multimodal analgesia.

Postoperative sternal wound pain will be judged by the Modified Objectice Pain Scale.

Postoperative sedation levels will be evaluated with Ramsya sedation score.

DETAILED DESCRIPTION:
Reducing the pain from surgical procedures performed early in life psychologically reduces the pain experienced by children in subsequent procedures. Pediatric cardiac surgery is associated with moderate to severe postoperative pain that is related to median sternotomy. Pediatric cardiac surgical patients usually undergo multiple surgical interventions and hospital admissions and will benefit from effective pain relief during their initial surgery. In a fast-track protocol, used in modern-day cardiac surgical care, early extubation may be facilitated by executive postoperative pain control, which also helps in maintaining hemodynamic stability.

Neuraxial analgesia techniques are eﬀective for sternotomy pain. However cardiac surgery procedures potentially require cardiopulmonary bypass (CPB) and systemic anticoagulation, thus increasing the epidural hematoma risk. Erector spinae plane (ESP) block appears to provide adequate regional analgesia for multiple dermatomal levels covering the sternum without increasing the risks associated with neuraxial blocks.

This prospective, randomized, and double-blind study is designed to examine the efficacy and safety of the ESP block on the postoperative analgesia in pediatric patients after cardiac surgery. We hypothesized that the ESP block significantly improves pain control, as evidenced by the reduced need for systemic postoperative analgesics.

METHOD After obtaining approval from the Institutional Review Boards at Çukurova University Medical Faculty, 40 pediatric patients aged 2-10 years, undergoing cardiac surgery with median sternotomy will be enrolled. Parental consent and patient assent from patients of an appropriate age will be obtained. Children with a preoperative ejection fraction<35%, a ventricular arrhythmia/dysrhythmia, a low cardiac output syndrome, a redo or an emergency surgery, a scoliosis or other anatomic contraindication to ESPB, a history of bleeding diathesis, an anticoagulant drug use at the time of the block and with known allergies to any of the study drugs will be excluded from the study.

Anesthesia Children received oral premedication of midazolam 0.5 mg/kg. After i.v. access will be obtained, fentanyl 5 µg/kg will be given. Anesthesia will be induced with 2-3 mg/kg propofol and all children will receive rocuronium 0,6 mg/kg for tracheal intubation. After tracheal intubation, an arterial line, central venous catheter, and urinary catheter will be inserted. Subsequently, fentanyl 5 µg/kg will be administered prior to incision and an additional 5 microg/kg of fentanyl given prior to CPB. Anesthesia will be maintained with %2-3 sevoflurane. Fentanyl 1 µg/kg will be given before skin closure at the end of surgery.

Intervention Patients were randomly assigned to a study group by the computer generated number table. Children in group B will be administered bilateral ESPB with 0.25% bupivacaine, while children in group C did not receive any intervention. The anesthesia resident observing the patient in the postperative period and the intensive care unit staff giving postoperative care will be blind to the study protocol.

Following anesthesia induction and endotracheal tube placement, the patient will be turned into a left lateral decubitus position and bilateral ESP block will be performed under aseptic conditions.

ESP block at bilateral side will be performed in the lateral decubitis position and at T5 transverse process level by using 10-MHz liner ultrasound probe. The probe will be located 1 cm lateral to T5 spinous process in longitudinal parasagittal orientation. Simplex A 50mm (B.Braun, Germany) will be inserted by using out of plane technique. The ESP blocks proceed with 0,5 ml/kg of 0,25% bupivacaine (Group B). The injection will be applied after the confirmation of location by hydrodissection developed anterior to erector spinae muscle with 1-2 ml of local anesthetic solution.

Postoperative care All the patients then will be shifted to the intensive care unit (ICU) after the surgery and managed with the institution's ICU protocol for postoperative pain management and ventilation.The postoperative analgesia will be provided with rescue intravenous (IV) morphine 0.05 mg/kg. Both the groups will receive IV paracetamol 15 mg/kg every 6 hours as a component of multimodal analgesia.

Postoperative sternal wound pain will be judged by the Modified Objectice Pain Scale.

Postoperative sedation levels will be evaluated with Ramsay sedation score.

ELIGIBILITY:
Inclusion Criteria:

* 2-10 years old patients
* Pediatric patients undergoing cardiac surgery with median sternotomy

Exclusion Criteria:

* A history of develop mental delay or mental retardation
* Any other heart defect
* Known allergy to any local anesthetic
* Clinically significant liver or renal disease.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours after arrival in Intensive care unit
  Total consumption of rescue analgesia by morphine (mcg/kg)

SECONDARY OUTCOMES:
Pain assesment in infant/toddlers | 24 hours after arrival in intensive care unit
  Pain assessment will be based on Modified objective pain scale

CONTACTS AND LOCATIONS:
Overall Officials: FERİDE KARACAER, Specialist, Principal Investigator — Cukurova University
Locations (1):
- Feri̇de Karacaer, Adana, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De la Cuadra-Fontaine JC, Concha M, Vuletin F, Arancibia H. Continuous Erector Spinae Plane block for thoracic surgery in a pediatric patient. Paediatr Anaesth. 2018 Jan;28(1):74-75. doi: 10.1111/pan.13277. No abstract available. PMID 29226529
- [Result] Barr AM, Tutungi E, Almeida AA. Parasternal intercostal block with ropivacaine for pain management after cardiac surgery: a double-blind, randomized, controlled trial. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):547-53. doi: 10.1053/j.jvca.2006.09.003. Epub 2006 Dec 22. PMID 17678782